CLINICAL TRIAL: NCT00228020
Title: A Randomized, Placebo-controlled, Double-blind, Multicenter Study Investigating Basiliximab in Combination With MMF, Cyclosporine Microemulsion and Prednisone in the Prevention of Acute Rejection in Pediatric Renal Allograft Recipients
Brief Title: Study of Safety and Efficacy of a Basiliximab, Mycophenolate Mofetil, Cyclosporine Microemulsion and Prednisone Combination Treatment Regimen in Pediatric Renal Allograft Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CCHI621ADE01
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2010-08

CONDITIONS: Pediatric Kidney Transplantation
Keywords: pediatric, kidney transplantation, basiliximab
MeSH Terms: interventions — Basiliximab; Cyclosporine; Prednisone; Steroids

ARMS (2):
- Basiliximab (Experimental): Patients will be on a regimen of Basiliximab, MMF, cyclosporine and steroids
  Interventions: Drug: basiliximab, MMF(mycophenolate mofetil), cyclosporine, prednisone (or equivalent)
- Basiliximab-free (Active Comparator): Patients will be on a regimen of MMF, cyclosporine and steroids.
  Interventions: Drug: MMF, cyclosporine, steroids

INTERVENTIONS:
Drug: basiliximab, MMF(mycophenolate mofetil), cyclosporine, prednisone (or equivalent)
  Arms: Basiliximab
Drug: MMF, cyclosporine, steroids
  Arms: Basiliximab-free

SUMMARY:
The aim of this study is assess the safety and efficacy of the treatment regimen of basiliximab ,cyclosporine microemulsion, MMF, and prednisone combined compared to cyclosporine microemulsion, MMF and prednisone in the time to first biopsy proven acute rejection episode or treatment failure during the first 6 months post-transplantation in pediatric renal allograft recipients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are recipients of primary or secondary renal allograft.
* Patients who are single-organ recipients (kidney only).

Exclusion Criteria:

•Patients who are recipients of HLA-identical renal transplants. Patients whose donor kidney cold ischemia time (CIT) is greater than 36 hours. Patients whose transplant kidney is obtained from a non-heart beating donor Other protocol-defined exclusion criteria may apply.

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Enrollment: 212 (Actual)
Dates: Start 2001-05; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Time to first BPAR episode or treatment failure | 6 months
  Treatment failure is defined as: graft loss, death, or initiation of anti-rejection therapy without prior biopsy-proven rejection (in case of medical contraindication for a biopsy).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis

REFERENCES:
- [Derived] Offner G, Toenshoff B, Hocker B, Krauss M, Bulla M, Cochat P, Fehrenbach H, Fischer W, Foulard M, Hoppe B, Hoyer PF, Jungraithmayr TC, Klaus G, Latta K, Leichter H, Mihatsch MJ, Misselwitz J, Montoya C, Muller-Wiefel DE, Neuhaus TJ, Pape L, Querfeld U, Plank C, Schwarke D, Wygoda S, Zimmerhackl LB. Efficacy and safety of basiliximab in pediatric renal transplant patients receiving cyclosporine, mycophenolate mofetil, and steroids. Transplantation. 2008 Nov 15;86(9):1241-8. doi: 10.1097/TP.0b013e318188af15. PMID 19005406
- [Derived] Hocker B, Kovarik JM, Daniel V, Opelz G, Fehrenbach H, Holder M, Hoppe B, Hoyer P, Jungraithmayr TC, Kopf-Shakib S, Laube GF, Muller-Wiefel DE, Offner G, Plank C, Schroder M, Weber LT, Zimmerhackl LB, Tonshoff B. Pharmacokinetics and immunodynamics of basiliximab in pediatric renal transplant recipients on mycophenolate mofetil comedication. Transplantation. 2008 Nov 15;86(9):1234-40. doi: 10.1097/TP.0b013e318188ae18. PMID 19005405